CLINICAL TRIAL: NCT00106405
Title: A Pilot Evaluation of the Safety and Efficacy of Memantine in Patients With Acute Mania Associated With Bipolar I Disorder
Brief Title: An Evaluation of the Safety and Efficacy of Memantine in Patients With Acute Mania Associated With Bipolar I Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: MEM-MD-27
Record Dates: First submitted 2005-03-24; First posted 2005-03-25 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Bipolar Disorder
Keywords: Bipolar I Disorder; Mania; Memantine HCl
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Memantine

INTERVENTIONS:
Drug: Memantine HCl

SUMMARY:
Bipolar disorder affects 2.4 million adults in the USA between the ages of 18-65 and has considerable economic impact on our society. Bipolar mania accounts for 1 in 7 psychiatric emergencies and is associated with significant morbidity and mortality. The purpose of the study is to evaluate the safety and efficacy of open-label memantine in the acute management of adults with bipolar I disorder hospitalized for mania.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a documented clinical diagnosis of bipolar I disorder and must be currently experiencing a manic or mixed episode.
* Patients must be voluntarily hospitalized with a primary diagnosis of mania.

Exclusion Criteria:

* Rapid cycling bipolar disorder.
* Suicidal risk.
* First manic episode.
* ECT, clozapine or a depot neuroleptic in the past 3 months.
* Substance dependence.
* Known HIV infection.
* Co-morbid serious, uncontrolled systemic illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-02; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Young Mania Rating Scale (YMRS)
Mania Rating Scale
Clinical Global Impression
Montgomery Asberg Depression Rating Scale
Positive and Negative Syndrome Scale (PANSS)
PANSS - Excited Component

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Synergy Clinical Research Center, National City, California
  - Sheppard Pratt Health System, Baltimore, Maryland
  - St. Charles Psychiatric Associates, Saint Charles, Missouri
  - Psychiatric Professional Services, Inc., Cincinnati, Ohio
  - Rebecca Sealy Hospital, Galveston, Texas
  - University Hills Clinical Research, Irving, Texas